CLINICAL TRIAL: NCT03863093
Title: Clinical Outcomes of Using Erythritol Powder by Means of Air Polishing With Ultrasonic Debridement in the Treatment of Initial Periodontal Pockets in Hand of Dental Students: A Split-mouth, Randomized, Comparative, Controlled Study
Brief Title: Evaluation of Air Polishing With Ultrasonic Debridement in the Treatment of Initial Periodontal Pockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syrian Private University (Other)
Responsible Party: Principal Investigator, Hala Albonni, Dr., Syrian Private University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SPU-DN-Perio-2
Record Dates: First submitted 2019-02-18; First posted 2019-03-05 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An erythritol powder (Experimental): An erythritol powder will be used by Electro Medical Systems AIRFLOW® and then Electro Medical Systems Piezo will be used for supra- and subgingival ultrasonic instrumentation
  Interventions: Device: Electro Medical Systems AIRFLOW®; Device: Electro Medical Systems Piezo
- ultrasonic instrumentation (Active Comparator): Electro Medical Systems Piezo will be used for supra- and subgingival ultrasonic instrumentation
  Interventions: Device: Electro Medical Systems Piezo

INTERVENTIONS:
Device: Electro Medical Systems AIRFLOW® — An erythritol powder will be used by Electro Medical Systems AIRFLOW® and then Electro Medical Systems Piezo will be used for supra- and subgingival ultrasonic instrumentation
  Arms: An erythritol powder
Device: Electro Medical Systems Piezo — Electro Medical Systems Piezo will be used for supra- and subgingival ultrasonic instrumentation

SUMMARY:
Clinical evaluation of using erythritol powder as air polishing with ultrasonic scaling and root planing in the treatment of initial periodontal pockets. This trial will be split-mouth design, in which each patient will receive traditional treatment (ultrasonic mechanical therapy and polishing) in one side, while the contralateral two quadrants of the jaws will be treated with erythritol powder by means of air polishing and ultrasonic scaling and root planing.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the usage of erythritol powder by means of air polishing in hand of undergraduate dental students as a single way to remove biofilm and the adjunctive application of ultrasonic piezo afterward for calculus removal and root planing only in the treatment of initial periodontal pockets.

The sample size will be 15 patients. Initially, oral hygiene instructions with scaling and root planing will consist of the treatment phase. Each subject will be informed comprehensively about oral hygiene instructions using disclosing solution (such as erythrosine) and hand mirror. The participant will be shown modified bass technique and the proper usage of dental floss and appropriate interdental brushes.

The control side will be treated with supra- and subgingival ultrasonic piezo scalers then supragingival polishing with rubber cup and a special fluoride containing paste as a traditional way of removal of plaque and calculus, while the test side, will be confined to erythritol powder by means of air polishing as the only way to remove ultrasonic piezo scalers.

At the end of treatment, hand instruments may be used to ensure the smoothness 0f the teeth surfaces.

Clinical measurements will be performed at baseline and at 2 weeks, 4 and 6 weeks for the plaque index and gingival indices, whereas probing will be performed only after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are in generally good health
2. Patients are from both gender and their age is between 18 to 60 years.
3. Patients have a minimum of 20 teeth
4. The patient is a non-smoker (less than 5 cigarettes per day) and non-alcoholic.
5. Female participants must not be pregnant or breastfeeding (lactation).
6. the absence of severe oral habits
7. the presence of at least one residual pocket with pocket depth >4 mm with interdental sites with a probing depth of 3 to 5 mm without furcation involvement or subgingival restorations.
8. A sign informed consent from participation and permission to use obtained data for research purposes.

Exclusion Criteria:

1. Bruxism
2. Allergy to glycine or chlorhexidine;
3. systemic medical conditions requiring antibiotic prophylaxis (for endocarditis prophylaxis) and anti-inflammatory drugs before dental procedures;
4. active systemic infectious disease;
5. major systemic illnesses (diabetes mellitus, cancer, immunodeficiency virus, bone metabolic diseases or disorders that compromise wound healing, radiation or immunosuppressive therapy, neutropenia, agranulocytosis, or bleeding disorders.
6. chronic high dose steroid therapy
7. Patients are undergone to radiotherapy or chemotherapy before or during the study period.
8. actively smoking more than five cigarettes per day;
9. signs of generalized severe periodontitis;
10. having received periodontal maintenance within 3 months before baseline
11. patients treated with antibiotics 6 months prior to the study
12. chronic bronchitis and asthma
13. compromised immune system
14. hypersensitivity to sugar alcohols.
15. any physical limitations or restrictions that might preclude normal oral hygiene procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-02-09 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
change in the papillary bleeding index | baseline, 2-weeks, 4-weeks, 6-weeks after the treatment
  Probing is performed in all four quadrants. A quadrant 1 is probed only from the oral aspect, quadrant 2 from the facial, 3 again from oral, and from the facial in quadrant 4
  Grade 1-Point: 20-30 seconds after probing the mesial and distal sulci with a periodontal probe, a single bleeding point is observed.
  Grade 2-Line/Points: A fine line of blood or several bleeding points become visible at the gingival margin.
  Grade 3-Triangle: The interdental triangle becomes more or less filled with blood.
  Grade 4-Drops: Profuse bleeding. Immediately after probing, blood flows into the interdental area to cover portions of the tooth and/or gingiva.
  Calculation:
  Papillary bleeding index= Bleeding Number/ Number of sites measured
change in the percentage of study sites positive for bleeding on probing | baseline, 6-weeks after the treatment
  All four surfaces of all teeth are assessed with regard to whether probing elicits bleeding (+) or not (-). The severity of gingivitis is expressed as a percentage.
  - no bleeding upon probing (not recorded)
  + bleeding upon probing
  Calculation:
  Bleeding on probing= Number of bleeding sites x100 / Number of sites evaluated

SECONDARY OUTCOMES:
change in the full mouth Plaque Index | baseline, 2-weeks, 4-weeks, 6-weeks after the treatment
  a score of 0 to 5 is assigned to each facial and lingual unrestored surface of all the teeth except third molars, as follows: The Plaque Index System
  Scores Criteria
  * 0 No plaque
  * 1 Separate flecks of plaque at the cervical margin of the tooth
  * 2 A thin continuous band of plaque (up to one mm) at the cervical margin of the tooth
  * 3 A band of plaque wider than one mm but covering less than one-third of the crown of the tooth
  * 4 Plaque covering at least one-third but less than two-thirds of the crown of the tooth
  * 5 Plaque covering two-thirds or more of the crown of the tooth
change in the Calculus index | baseline, 2-weeks, 4-weeks, 6-weeks after the treatment
  * 0, no calculus;
  * 1, mild supragingival calculus extending to marginal gingiva is present;
  * 2, moderate supra and subgingival calculus or only subgingival calculus is present; and
  * 3, excessive supra and subgingival calculus is present.
  it will be estimated visually
change in the Modified Gingival Index | baseline, 2-weeks, 4-weeks, 6-weeks after the treatment
  * 0 = Normal gingiva;
  * 1 = Mild inflammation - slight change in color and slight edema;
  * 2 = Moderate inflammation - redness, edema and glazing;
  * 3 = Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.
  it will be estimated visually
change in the Probing pocket depth | baseline, 6- weeks after the treatment
  measure as the change in distance from the gingival margin to the bottom of the gingival sulcus by using a periodontal probe (UNC 15 "University of North Carolina")
The change of the root sensitivity | baseline, 24- hours, 48- hours, 72-hours, 1- week, 2-weeks, 4-weeks, 6-weeks after the treatment
  will be evaluated using a visual analogue scale (VAS). The VAS root sensitivity scores ranges between 0 to 10. (0: no root sensitivity, 5: moderate root sensitivity, 10: severe root sensitivity).

CONTACTS AND LOCATIONS:
Overall Officials: Hala Albonni, DDS MSc, Principal Investigator — Syrian Private University; Hazem Sawaf, DDS MSc PhD, Study Chair — Syrian Private University
Locations (1):
- Syrian Private University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flemmig TF, Arushanov D, Daubert D, Rothen M, Mueller G, Leroux BG. Randomized controlled trial assessing efficacy and safety of glycine powder air polishing in moderate-to-deep periodontal pockets. J Periodontol. 2012 Apr;83(4):444-52. doi: 10.1902/jop.2011.110367. Epub 2011 Aug 23. PMID 21861637
- [Background] Hagi TT, Hofmanner P, Salvi GE, Ramseier CA, Sculean A. Clinical outcomes following subgingival application of a novel erythritol powder by means of air polishing in supportive periodontal therapy: a randomized, controlled clinical study. Quintessence Int. 2013 Nov-Dec;44(10):753-61. doi: 10.3290/j.qi.a30606. PMID 24078975
- [Background] Muller N, Moene R, Cancela JA, Mombelli A. Subgingival air-polishing with erythritol during periodontal maintenance: randomized clinical trial of twelve months. J Clin Periodontol. 2014 Sep;41(9):883-9. doi: 10.1111/jcpe.12289. Epub 2014 Aug 7. PMID 25041441
- [Background] Moene R, Decaillet F, Andersen E, Mombelli A. Subgingival plaque removal using a new air-polishing device. J Periodontol. 2010 Jan;81(1):79-88. doi: 10.1902/jop.2009.090394. PMID 20059420
- [Background] Park EJ, Kwon EY, Kim HJ, Lee JY, Choi J, Joo JY. Clinical and microbiological effects of the supplementary use of an erythritol powder air-polishing device in non-surgical periodontal therapy: a randomized clinical trial. J Periodontal Implant Sci. 2018 Oct 24;48(5):295-304. doi: 10.5051/jpis.2018.48.5.295. eCollection 2018 Oct. PMID 30405937
- [Background] Wennstrom JL, Dahlen G, Ramberg P. Subgingival debridement of periodontal pockets by air polishing in comparison with ultrasonic instrumentation during maintenance therapy. J Clin Periodontol. 2011 Sep;38(9):820-7. doi: 10.1111/j.1600-051X.2011.01751.x. Epub 2011 Jul 7. PMID 21736599